CLINICAL TRIAL: NCT05521958
Title: Genetics and Local Gene Expression in Lower Extremity Acute Traumatic Compartment Syndrome
Brief Title: Gene Expression in Lower Extremity Acute Traumatic Compartment Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, Principle Investigator, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 152310
Record Dates: First submitted 2022-08-15; First posted 2022-08-30 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Tibial Shaft Fracture; Tibial Plateau Fracture
Keywords: tibial shaft or tibial plateau fracture; acute compartment syndrome; without acute compartment syndrome; exertional compartment syndrome; gene expression; myostatin
MeSH Terms: conditions — Tibial Plateau Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acute tibial shaft or tibial plateau fractures without compartment syndrome (Other): Patients with acute lower leg fractures who do not have clinical compartment syndrome.
  Interventions: Procedure: Acute injury without compartment syndrome
- Acute tibial shaft or tibial plateau fractures with compartment syndrome. (Other): Patients with acute lower leg fractures with acute compartment syndrome.
  Interventions: Procedure: Acute injury with compartment syndrome
- Exertional compartment syndrome (Other): Patients with a diagnosis of exertional compartment syndrome who are planning to undergo surgical procedure to release the compartment fascia will be recruited to participate prior to surgical intervention.
  Interventions: Procedure: Exertional compartment syndrome

INTERVENTIONS:
Procedure: Acute injury without compartment syndrome — Acute tibial shaft or tibial plateau fractures who do not have clinical compartment syndrome.
  Muscle punch biopsy of the anterior compartment will be taken.
  Arms: Acute tibial shaft or tibial plateau fractures without compartment syndrome
Procedure: Acute injury with compartment syndrome — Acute tibial shaft or tibial plateau fractures who have clinical compartment syndrome.
  Muscle punch biopsy of the anterior compartment will be taken.
  Arms: Acute tibial shaft or tibial plateau fractures with compartment syndrome.
Procedure: Exertional compartment syndrome — For patients with exertional compartment syndrome, a muscle biopsy will be obtained from affected extremity.
  Arms: Exertional compartment syndrome

SUMMARY:
The purpose of this study is to evaluate both genotypic differences and differences in local gene expression in individuals who develop acute traumatic compartment syndrome relative to control patients with at-risk lower extremity fractures who do not develop compartment syndrome.

DETAILED DESCRIPTION:
Acute compartment syndrome is associated with infection, contractures, fracture non-union, and chronic pain syndromes. The most common cause of acute compartment syndrome is fracture. Individuals with compartment syndrome associated with a lower extremity fracture have demonstrated worse patient reported outcome scores compared to individuals who suffer lower extremity fractures alone.

The pathophysiology of compartment syndrome has been traditionally described as loss of tissue perfusion and subsequent cellular anoxia related to supra-physiologic pressure within a closed myofascial space. Both animal and clinical studies have suggested that compartment syndrome develops when the intra-compartmental pressure approaches systemic diastolic blood pressure. However, other studies have demonstrated that high absolute compartment pressures and/or narrowed delta pressures have poor sensitivity for predicting compartment syndrome, suggesting that the pathophysiology of compartment syndrome is likely more complex than the currently accepted understanding of the disease process.

Animal models suggest that fracture promotes inflammation and exacerbates microvascular dysfunction, which may act synergistically with elevated intra-compartmental pressures to create clinical compartment syndrome. It is known that fracture causes microvascular damage and inflammation in surrounding muscle tissue. Several models have demonstrated that the microvascular environment in compartment syndrome is characterized by tenuous, intermittent blood supply to the musculature, which displays asymmetric microvascular dysfunction in response to elevated compartment pressures. Similarly, recent animal research has demonstrated that elevated intra-compartmental pressure is associated with a pro-inflammatory state, which directly contributes to skeletal muscle injury and may exacerbate microvascular injury.

It is unknown whether individual genomic and/or transcriptomic variability is clinically relevant with respect to response to fracture or the development of compartment syndrome. However, there is evidence from the vascular surgery literature in both animal and human models that individual variability in gene expression meaningfully affects skeletal muscle response to acute ischemia. The investigators hypothesize that there may be an individual pre-disposition to developing clinical compartment syndrome in the setting of at-risk fractures which manifests itself in the cellular response to inflammation and low grade ischemia. The overarching goal of this study is to characterize cellular level dysfunction in human compartment syndrome and to determine whether there are unique gene expression profiles associated with the development of clinical compartment syndrome. Specific aim 1 of this study is to compare genetic and transcriptomic differences individuals with high-risk tibia fractures who do not develop compartment syndrome and individuals with high-risk tibia fractures who do develop clinical compartment syndrome. Specific aim 2 of this study is to to compare genetic differences between acute compartment syndrome patients and chronic exertional compartment syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18+ years of age. English speaking.
* Patients with the clinical diagnosis of lower leg acute compartment syndrome secondary to tibial shaft or tibial plateau fracture.
* Patients without clinical compartment syndrome undergoing operative intervention within 48 hours of injury for tibial shaft or tibial plateau fractures.
* Patients with the clinical diagnosis of exertional compartment syndrome with planned surgical intervention.

Exclusion Criteria:

* Non-english speaking participants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Myostatin (% increase) | Immediately after the muscle tissue harvest procedure.
  The investigators primary marker of interest is myostatin. The investigators will determine the (%) increase in myostatin levels in muscle tissues between compartment syndrome patients versus fracture controls. (%) increase in myostatin levels in muscle tissues between compartment syndrome patients versus patients with exertional compartment syndrome will also be determined. The measurement tool is polymerase chain reaction (PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No